CLINICAL TRIAL: NCT04345978
Title: Effects of Different Fasting Strategies in Perioperative Period on Postoperative Recovery, Immune Function, and Long-term Prognosis in Patients With Radical Resection of Colorectal Cancer
Brief Title: Effects of Fasting Strategies on Postoperative Recovery and Long-term Prognosis in Patients With Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Cancer Hospital, China (Other); Huashan Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tongji Hospital (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Changhong Miao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2020-063
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Fasting; Immune Suppression; Complication of Surgical Procedure; Colorectal Cancer
Keywords: Fasting; Immune Suppression; Survival; Immune metabolism
MeSH Terms: conditions — Fasting; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Fasting (Placebo Comparator): The patient starts fasting 8 hours before the operation,and does not take any solid or liquid foods and nutrients during the fasting process.The fasting period does not strictly limit the consumption of pure water,After surgery 8 hours,the patients was allowed to feeding.
  Interventions: Behavioral: Fasting hours
- Prolong Fasting (Experimental): The patient starts fasting 24 hours before the operation, and does not take any solid or liquid foods and nutrients during the fasting process. The fasting period does not strictly limit the consumption of pure water.After surgery 24 hours,the patients was allowed to feeding.
  Interventions: Behavioral: Fasting hours

INTERVENTIONS:
Behavioral: Fasting hours — Normal Fasting hours before CRC surgery for 8 hours and feeding 8 hours after surgery; Prolong fasting hours before CRC surgery for 24 hours and feeding 24 hours after surgery.

SUMMARY:
In 2018, colorectal cancer is the third most common malignant tumor in terms of morbidity and second mortality in the world. Surgical resection is still the main treatment for colorectal cancer.With the introduction of the ERAS, the latest international and domestic guidelines for fasting before surgery all advocate shortening the fasting time. For example, 2 hours before surgery, oral take cleared fluids, including water, sugar water, fruit juice, tea and black coffee (without milk) is allowed.Solid food can be consumed 4 hours before surgery, and oral diet should be resumed as soon as possible after surgery. Changes in diet, nutritional status, and physical activity are closely related to the incidence of colorectal cancer. Therefore, we believe that the intestine may be very sensitive to different fasting times during the perioperative period. Prolonging the fasting time may improve the prognosis by improving postoperative insulin resistance, reducing inflammation and protecting anti-tumor immune function in patients with colorectal cancer.Prolonged fasting time seems to be contrary to the results of some studies, and whether it is applicable to patients with tumor surgery is unclear. Therefore, there is an urgent need to conduct large-scale, prospective, randomized controlled clinical studies to clarify the most suitable perioperative fasting strategy (including composition, interval, and amount) for cancer patients, which can not only reduce surgical stress and speed up postoperative rehabilitation,reduce postoperative metastasis and recurrence and improve mid- and long-term prognosis.

DETAILED DESCRIPTION:
As early as a century ago, Investigators proved that diet restriction can prevent the occurrence of transplanted tumors in mice. Following this milestone, many animal studies (from mice to primates) have confirmed that diet restriction can slow the development of spontaneous tumors and transplanted tumors. A study of macaque monkeys for more than 20 years revealed that restricting diet by 30% can reduce the incidence of tumors by 50%, which makes people see the potential value of restricting diet to humans. However, whether diet restriction can also reduce the incidence of human tumors is not entirely clear. The growth of tumor cells requires a nutrient-rich environment, and the lack of glucose and amino acids caused by diet restrictions is very detrimental to tumor cells. Unlike normal cells, tumor cells mainly rely on glycolysis (Warburg effect) rather than energy and biosynthetic precursors provided by oxidative phosphorylation for proliferation. These characteristics make tumor cells extremely sensitive to changes in the surrounding environment, which is called differential stress sensitization (DSS).Investigators found that the use of low sugar and low serum in a cell model to simulate periodic fasting can enhance the sensitivity of human or animal tumor cells to doxorubicin and cyclophosphamide, and also found that they were transplanted subcutaneously in mice Melanoma or breast cancer, diet combined with chemotherapy is better than chemotherapy alone; in the mouse metastatic neuroblastoma model, fasting before high-dose chemotherapy can successfully reduce the toxic side effects of chemotherapy drugs and reduce metastasis and prolong the tumor-free survival. Surgery and stress are twin brothers. Surgical resection, blood flow blockage, ischemia-reperfusion injury, tissue damage, local inflammatory factor release, and changes in systemic neuroendocrine and metabolism all affect blood flow, blood coagulation, and immune function. Investgators found restricted diet can reduce the inflammatory response after myocardial ischemia-reperfusion injury in mice. Many animal experiments have confirmed that perioperative fasting can effectively protect the liver, kidneys, and brain from organ damage. The specific mechanism may be related to fasting increasing antioxidant enzyme activity, reducing insulin-like growth factor-1 (IGF-1), and activating the autophagy pathway. Similar to chemotherapy, there is currently no randomized clinical controlled study to evaluate the impact of individualized perioperative dietary regimens (such as restricted diet) on the prognosis of tumor surgery.

In 2018, colorectal cancer is the third most common malignant tumor in terms of morbidity and second mortality in the world. Surgical resection is still the main treatment for colorectal cancer.With the introduction of the ERAS, the latest international and domestic guidelines for fasting before surgery all advocate shortening the fasting time. For example, 2 hours before surgery, oral take cleared fluids, including water, sugar water, fruit juice, tea and black coffee (without milk) is allowed.Solid food can be consumed 6 hours before surgery, and oral diet should be resumed as soon as possible after surgery. Changes in diet, nutritional status, and physical activity are closely related to the incidence of colorectal cancer. Therefore, we believe that the intestine may be very sensitive to different fasting times during the perioperative period. Prolonging the fasting time may improve the prognosis by improving postoperative insulin resistance, reducing inflammation and protecting anti-tumor immune function in patients with colorectal cancer.Prolonged fasting time seems to be contrary to the results of some studies, and whether it is applicable to patients with tumor surgery is unclear. Therefore, there is an urgent need to conduct large-scale, prospective, randomized controlled clinical studies to clarify the most suitable perioperative fasting strategy (including composition, interval, and amount) for cancer patients, which can not only reduce surgical stress and speed up postoperative rehabilitation,reduce postoperative metastasis and recurrence and improve mid- and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 ~ 70 years old
2. With BMI 20.5-25.0 kg/m2
3. Without any Endocrine and metabolic diseases
4. A stable body weight (±3 kg) for at least 6 months
5. Those diagnosed with colorectal cancer by preoperative pathology or enteroscopy
6. Patients undergoing laparoscopic radical colorectal cancer resection
7. ASA grade I-III grade
8. Initial patients have not received any treatment for bowel cancer except neoadjuvant chemotherapy
9. Patients with confirmed and feasible radical resection of colorectal cancer
10. No evidence of distant metastasis before surgery
11. Willing to participate in the research of the subject and agree to follow up regularly

Exclusion Criteria:

1. Patients with relapsed colorectal cancer who are going to undergo surgery and re-excision
2. accompanied by other malignant tumors
3. Severe malnourished patients
4. History of systemic metabolism such as diabetes
5. Before surgery, have received other treatments for colorectal cancer (such as local excision, etc.) in addition to neoadjuvant chemotherapy
6. Have a history of immunotherapy before surgery
7. Combined with basic diseases of serious heart, lung, brain, kidney and other important organs
8. Combined with severe primary diseases such as severe immune system or hematopoietic system
9. The tumor burden cannot be cured, and there is distant metastasis. Those who intend to undergo palliative surgery
10. People with gastroesophageal reflux disease, difficulty swallowing, intestinal obstruction, or difficulty in airway management
11. People who refuse to participate in the study or cannot receive long-term follow-up

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | During 2 years after surgery
  Defined and calculated as the time from the date of surgery to the first time of colon cancer recurrence or metastasis or cancer-related death

SECONDARY OUTCOMES:
Overall Survival | During 2 years after surgery
  Defined and calculated as the time from the date of surgery to the first time of Colon cancer recurrence or metastasis or cancer-related death
Postoperative pain score and side effects of patient-controlled analgesia | During the first 48 hours after surgery
  Assessed with visual analogue score ( 0 is no pain and 10 is the most severe pain)
Incidence of delirium | During the first 1 week after surgery
  Assessed for delirium using the 3D-CAM instrument
Length of stay in hospital after surgery and total costs after surgery | During the first 30 days after surgery
  Length of stay in hospital after surgery and total costs after surgery
Return of bowel function | During the first 30 days after surgery
  Measured by the time of first flatus
Neutrophil to Lymphocyte Ratio，LMR,SII | During the first24、48 and 72 hours after surgery
  Neutrophil to Lymphocyte Ratio,Lymphocyte to Monocyte ratio,Symstem Imflammatory Index
Serum CA19-9 、CA125、CEA、CA72-4、CA242、AFP、CA15-3、CA50 levels | During 2 years after surgery
  Tumor Biomaker Level
Recovery Parameter | During the first24、48 and 72 hours after surgery
  Q40 scale score
T Lymphocyte cell count | During the first24、48 and 72 hours after surgery
  T lymphocyte cell count before fasting and after fasting
T Lymphocyte cell DNA damage | During the first24、48 and 72 hours after surgery
  T lymphocyte cell count before fasting and after fasting
IL-1β，IL-2,IL-4,IL-5,IL-6,IL-8,IL-10,IL-17A,IL-17F,TNF-α，TNF-β， | During the first24、48 and 72 hours after surgery
  Inflammatory factor level

CONTACTS AND LOCATIONS:
Overall Officials: Mengjie Yang, phD, Principal Investigator — Fudan University
Locations (7):
- China (7):
  - Department of Biostatistics, School of Public Health, Fudan University,, Shanghai, Shanghai Municipality
  - Fudan University Huashan Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer center, Shanghai, Shanghai Municipality
  - Fudan University,ZhongShan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Naval Medical University,, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital,Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital,Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No